CLINICAL TRIAL: NCT04101864
Title: Electromagnetic Navigation System Versus Freehand Technique in Total Hip Arthroplasty: A Prospective Randomized Study
Brief Title: Electromagnetic Navigation System Versus Freehand Technique in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valdoltra Orthopedic Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77/05/12
Record Dates: First submitted 2019-09-09; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Hip Osteoarthritis
Keywords: navigation; hip arthroplasty; surgical time; landmark
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Sample size will be calculated. The Consolidated Standards of Reporting Trials statement guidelines will be followed to perform this prospective, randomized, controlled, trial and to present the results. Included patients will be randomly allocated in a 1:1 ratio into the study and the control group. Randomization will be conducted using computer-generated numbers.
Who Masked: Outcomes Assessor
Masking Description: Postoperative computed tomography measurements of acetabular component position will be done by independent technician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromagnetic navigation (Experimental): In the study group acetabular components in total hip arthroplasty will be placed with the help of electromagnetic image-less navigation system. Reference plane will be anterior pelvic plane.
  Interventions: Procedure: Electromagnetic navigation
- Freehand (Active Comparator): In the control group acetabular components in total hip arthroplasty will be placed with the help of the freehand technique.
  Interventions: Procedure: Freehand

INTERVENTIONS:
Procedure: Electromagnetic navigation — Acetabular component placement in total hip arthroplasty will be performed wit the help of electromagnetic image-less navigation system.
  Arms: Electromagnetic navigation
Procedure: Freehand — In the control group acetabular components in total hip arthroplasty will be placed with the help of the freehand technique.
  Arms: Freehand

SUMMARY:
A prospective randomized study comparing accuracy and precision of acetabular component placement in total hip arthroplasty with use of novel electromagnetic navigation system versus freehand technique.

DETAILED DESCRIPTION:
Patients with hip arthritis, who are to be treated with total hip arthroplasty will be randomized in two groups. Patents allocated to study group will get their acetabular components implanted with the help of electromagnetic navigation system. Patients allocated to the control group will get their acetabular components implanted with freehand technique. Accuracy and precision of implanted acetabular components will be assessed on images obtained by postoperative computed tomography. Postoperative inclination and anteversion angles of acetabular components will be measured by the independent technician. Results will be statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* unilateral surgery
* osteoarthritis of the hip
* no previous surgery on the affected hip
* implantation of the same acetabular component through the same approach
* signed informed consent

Exclusion Criteria:

* age under 18 years
* unwilling to participate
* prior surgery on affected hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Acetabular component position | Up to 48 hours after surgery
  Comparison of the precision and the accuracy of acetabular components between both groups

SECONDARY OUTCOMES:
Surgical time | Immediately after surgical procedure
  Comparison of duration of surgery between both groups
Clinical result | 8-10 weeks postoperatively
  Comparison of improvement of Harris hip score between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Rene Mihalič, MD, Principal Investigator — Valdoltra Orthopedic Hospital; Rihard Trebše, MD, PhD, Study Director — Valdoltra Orthopedic Hospital
Locations (1):
- Valdoltra Orthopedic Hospital, Ankaran, Slovenia

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.